CLINICAL TRIAL: NCT06694285
Title: Observational Study on the Role of Chest Ultrasound in Patients With Respiratory Tract Infections
Brief Title: The Role of Chest Ultrasound in Patients With Respiratory Tract Infections
Acronym: REPSECO
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6520
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-11

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound evaluation — The subjects will constitute a cohort whose medical history, clinical, ultrasound and treatment data reported in the appropriate data collection form will be prospectively collected. Enrolled patients will undergo clinical and ultrasonographic evaluation in a manner not unlike routine clinical practice.

SUMMARY:
Respiratory tract infections are a major cause of hospitalization among pediatric and adult patients, regardless of the cause, whether viral or bacterial. It is critical to stratify each patient's risk to predict the subsequent clinical course. Point-of-care chest ultrasonography in parallel with clinical evaluation has been found to be an effective tool to assess the severity of pathology. A number of scores have been validated on the basis of the ultrasound picture. Currently, a growing interest is directed toward the unambiguous validation of an ultrasound score that can predict the patient's outcome in terms of hospitalization, ICU admission, need for a more pronounced approach in terms of respiratory care both qualitatively and quantitatively.

DETAILED DESCRIPTION:
Acute respiratory infections are the leading cause of illness and mortality in children under five, with children experiencing three to six episodes annually. This prevalence remains consistent across various demographics, although the severity of these infections differs significantly between high- and low-income countries. In developing nations, factors such as specific pathogens and risk factors contribute to higher mortality rates from these diseases. The most common respiratory infections in young children include pneumonia and bronchiolitis. Bronchiolitis, primarily caused by respiratory syncytial virus (RSV), is a significant viral infection affecting infants, particularly those under one year old, with peak incidence between three to six months. RSV affects 50-80% of bronchiolitis cases, while other viruses like rhinoviruses and influenza may also play roles. The American Academy of Pediatrics recommends a clinical diagnosis for bronchiolitis, reserving chest radiography for severe cases to exclude other conditions. Treatment is largely supportive, focusing on hydration and respiratory care, with only about 6% of cases requiring intensive care unit admission. Bacterial pneumonia is another major respiratory infection in children, often caused by Streptococcus pneumoniae or Haemophilus influenzae type b (Hib). Atypical pneumonias can arise from Mycoplasma pneumoniae and Chlamydia pneumoniae, particularly in older children. Current guidelines suggest that patients with uncomplicated community-acquired pneumonia do not require chest imaging or laboratory tests and can often be treated at home. Effective clinical assessment is crucial for stratifying risk in respiratory infections. Vital signs such as heart rate and respiratory rate, along with physical examination findings like wheezing or use of accessory muscles, help predict clinical outcomes. However, these assessments can be complicated by factors like fever or patient compliance issues. Recent studies have highlighted the utility of lung ultrasonography as a point-of-care tool for assessing various pulmonary conditions in pediatrics, correlating ultrasound patterns with disease severity. In pediatric acute respiratory distress syndrome (PARDS), a new definition has emerged that shifts focus from bilateral infiltrates to the saturation-to-inhaled oxygen fraction (S/F) ratio for assessing severity. An S/F ratio below 235 indicates moderate PARDS, while below 212 signifies severe PARDS. This approach enhances the evaluation of respiratory distress in children, providing a more practical method for predicting clinical outcomes based on easily obtainable parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0 to 20 years with a clinical diagnosis of respiratory tract infection, evaluated in the emergency department and then discharged home or admitted to the Pediatric Intensive Care Unit or Pediatrics Department.
* Informed consent signed by parents or patient of legal age

Exclusion Criteria:

* Refusal to sign informed consent
* Patients with bronchopulmonary dysplasia
* Foreign body aspiration cases
* Patients with pulmonary malformations
* Patients with neuromuscular diseases
* Patients with hemodynamically significant congenital heart disease

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 0 to 20 years with a clinical diagnosis of respiratory tract infection, evaluated in the emergency department and then discharged home or admitted to the Pediatric Intensive Care Unit or Pediatrics Department.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
The ultrasound pattern of patients with respiratory tract infections | 1 hour
  To evaluate the ultrasound pattern of patients with respiratory tract infections by score.

SECONDARY OUTCOMES:
the duration of hospitalization | 1 hour
  Validate a qualitative and quantitative ultrasound protocol to assess respiratory tract infections to predict the duration of hospitalization
Use the SatO2/FiO2 ratio to evaluate outcome | 20 minutes
  Use the SatO2/FiO2 ratio in conjunction with clinical assessment to evaluate the initiation of respiratory assistance with high-flow oxygen
correlation between ultrasound score and vital parameters | 1 hour
  Assess a correlation between ultrasound score and vital parameters (FR, HR, SatO2)
correlation between ultrasound score and indices of inflammation | 1 hour
  Assess a correlation between ultrasound score and indices of inflammation (PCR, PCT)
correlation between ultrasound parameters and etiology | 2 days
  Evaluate a possible correlation between ultrasound parameters (paravertebral consolidations, multiple confluent B-lines, white lung) and etiology (positive virus swab for VRS or other respiratory viruses)
possible correlations between various epidemiologic and clinical data | 2 hours
  Assess possible correlations between various epidemiologic and clinical data of patients with respiratory tract infections, collected retrospectively over the past 10 years at the Pediatric Emergency Department in order to analyze trends of different etiologic agents and age groups affected with the aim of having useful data for planning prevention strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gatto, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS UOSD Pronto Soccorso Pediatrico, Rome, Lazio, Italy